CLINICAL TRIAL: NCT03267667
Title: Effect of Obstructive Sleep Apnea on Right Ventricle Heamodynamics and Function
Brief Title: Effect of OSA on RV Heamodynamics and Function
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mary Zakher Bakhiet, resident doctor, Assiut University
Other Study IDs: 17100300
Record Dates: First submitted 2017-08-25; First posted 2017-08-30 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Sleep Apnea, Obstructive
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- obstructive sleep apnea patients: number of 90 patients will be investigated by 2D echocardiography and cardiac MRI to determine the right ventricle function
  Interventions: Diagnostic Test: 2D Echocardiography and cardiac MRI
- healthy volunteers: number of 10 subjects will be investigated by 2D echocardiography and cardiac MRI to determine right ventricular function in healthy persons have risk factors other than cardiac or lung diseases
  Interventions: Diagnostic Test: 2D Echocardiography and cardiac MRI

INTERVENTIONS:
Diagnostic Test: 2D Echocardiography and cardiac MRI — imaging of right ventricle by both modalities to assess right ventricle function accurately

SUMMARY:
Correlation of severity of obstructive sleep apnea and function of the right ventricle by means of 2D echocardiography and cardiac MRI

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a frequently under diagnosed condition that has emerged as an increasing medical problem with important social and financial implications worldwide. OSA is a well established risk factor for systemic hypertension , myocardial infarction or stroke.

Obstructive sleep apnea syndrome (OSAS) is characterized by repetitive collapse of the upper airway during sleep .The obstructive apneic event is associated with considerable breathing efforts against a totally or partially occluded upper airway, and apnea is terminated by an arousal and heavy snoring as airflow is restored. Severity of OSAS is described according to total number of apneas and hyperpneas per hour of sleep, which is named as the apnea-hypopnea index (AHI).

Cardiovascular disturbances are the most serious complications of OSAS. These complications include heart failure, acute myocardial infarction, nocturnal arrhythmias, stroke, systemic and pulmonary hypertension. All these cardiovascular complications increase morbidity and mortality of OSAS.

Currently, sleep apnea is accepted as one of the identifiable causes of hypertension. Also, OSAS is closely associated with obesity and ageing.

There is conclusive evidence that OSAS influences right heart function (the pathophysiological consequences of sleep apnea-hypopnea might result in an imbalance in myocardial oxygen delivery/consumption ratio, activation of sympathetic and other neurohormonal systems, and increased right and left ventricular after load )

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed as OSA with age range from 18 to 70 years
* Glomerular filtration rate (MDRD formula-based) > 60 ml/min
* Arterial hypertension diagnosed according to the European Society of Hypertension 2013 Guidelines.

Exclusion Criteria:

* Mental illness
* Acute and chronic inflammation
* Heart failure III or IV grade
* Chronic administration of drugs with confirmed nephrotoxicity and/or sympathicomimetics
* Obstructive and restrictive pulmonary diseases which may deteriorate the function of the respiratory system

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will include 90 patients who are diagnosed as obstructive sleep apnea by sleep study and 10 healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
The RV function in subjects with OSA compared with healthy persons | 1 year
  Assessment of RV function by cardiac MRI in OSA patients and healthy volunteers

SECONDARY OUTCOMES:
Early detection of any impairment in cardiac global function in the participants before causing symptoms. | 1 year
  Cardiac MRI help to detect early cardiac dysfunction before symptoms appear which causes. Early detection equal early management which will improve the cardiac prognosis

CONTACTS AND LOCATIONS:
Overall Officials: Salwa R. Demitry, Study Director — Assiut University; Aliaë A. Mohamid, Study Director — Assiut University; Ayman k. Hassan, Study Director — Assiut University
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nieto FJ, Young TB, Lind BK, Shahar E, Samet JM, Redline S, D'Agostino RB, Newman AB, Lebowitz MD, Pickering TG. Association of sleep-disordered breathing, sleep apnea, and hypertension in a large community-based study. Sleep Heart Health Study. JAMA. 2000 Apr 12;283(14):1829-36. doi: 10.1001/jama.283.14.1829. PMID 10770144
- [Background] Peppard PE, Young T, Palta M, Skatrud J. Prospective study of the association between sleep-disordered breathing and hypertension. N Engl J Med. 2000 May 11;342(19):1378-84. doi: 10.1056/NEJM200005113421901. PMID 10805822
- [Background] Hung J, Whitford EG, Parsons RW, Hillman DR. Association of sleep apnoea with myocardial infarction in men. Lancet. 1990 Aug 4;336(8710):261-4. doi: 10.1016/0140-6736(90)91799-g. PMID 1973968
- [Background] Palomaki H, Partinen M, Erkinjuntti T, Kaste M. Snoring, sleep apnea syndrome, and stroke. Neurology. 1992 Jul;42(7 Suppl 6):75-81; discussion 82. PMID 1630643
- [Background] Guilleminault C, Tilkian A, Dement WC. The sleep apnea syndromes. Annu Rev Med. 1976;27:465-84. doi: 10.1146/annurev.me.27.020176.002341. No abstract available. PMID 180875
- [Background] Lattimore JD, Celermajer DS, Wilcox I. Obstructive sleep apnea and cardiovascular disease. J Am Coll Cardiol. 2003 May 7;41(9):1429-37. doi: 10.1016/s0735-1097(03)00184-0. PMID 12742277
- [Background] Malone S, Liu PP, Holloway R, Rutherford R, Xie A, Bradley TD. Obstructive sleep apnoea in patients with dilated cardiomyopathy: effects of continuous positive airway pressure. Lancet. 1991 Dec 14;338(8781):1480-4. doi: 10.1016/0140-6736(91)92299-h. PMID 1683918
- [Background] Guilleminault C, Connolly SJ, Winkle RA. Cardiac arrhythmia and conduction disturbances during sleep in 400 patients with sleep apnea syndrome. Am J Cardiol. 1983 Sep 1;52(5):490-4. doi: 10.1016/0002-9149(83)90013-9. PMID 6193700
- [Background] Weitzenblum E, Krieger J, Apprill M, Vallee E, Ehrhart M, Ratomaharo J, Oswald M, Kurtz D. Daytime pulmonary hypertension in patients with obstructive sleep apnea syndrome. Am Rev Respir Dis. 1988 Aug;138(2):345-9. doi: 10.1164/ajrccm/138.2.345. PMID 3143285
- [Background] Chobanian AV, Bakris GL, Black HR, Cushman WC, Green LA, Izzo JL Jr, Jones DW, Materson BJ, Oparil S, Wright JT Jr, Roccella EJ; National Heart, Lung, and Blood Institute Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure; National High Blood Pressure Education Program Coordinating Committee. The Seventh Report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure: the JNC 7 report. JAMA. 2003 May 21;289(19):2560-72. doi: 10.1001/jama.289.19.2560. Epub 2003 May 14. PMID 12748199
- [Background] Levinson PD, McGarvey ST, Carlisle CC, Eveloff SE, Herbert PN, Millman RP. Adiposity and cardiovascular risk factors in men with obstructive sleep apnea. Chest. 1993 May;103(5):1336-42. doi: 10.1378/chest.103.5.1336. PMID 8486007
- [Background] Ancoli-Israel S, Coy T. Are breathing disturbances in elderly equivalent to sleep apnea syndrome? Sleep. 1994 Feb;17(1):77-83. doi: 10.1093/sleep/17.1.77. No abstract available. PMID 8191206
- [Background] Javaheri S. Central sleep apnea in congestive heart failure: prevalence, mechanisms, impact, and therapeutic options. Semin Respir Crit Care Med. 2005 Feb;26(1):44-55. doi: 10.1055/s-2005-864206. PMID 16052417